CLINICAL TRIAL: NCT07117071
Title: Prevalence of Fuchs Endothelial Corneal Dystrophy in a Population of Dermatology Patients.
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN1392025/CHUSTE
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Fuchs Endothelial Corneal Dystrophy
Keywords: Fuchs endothelial corneal dystrophy; specular microscopy; prevalence; carcinoma
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy; Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- screening of Fuchs endothelial corneal dystrophy: Patients with screening of Fuchs endothelial corneal dystrophy will be included.
  Interventions: Other: collection of medical data

INTERVENTIONS:
Other: collection of medical data — collection of medical data : Age, Sex, Previous cataract surgery, Cellularity, Dermatological pathology, results of screening of Fuchs endothelial corneal dystrophy by Specular microscopy

SUMMARY:
The prevalence of Fuchs Endothelial Corneal Dystrophy (FECD) varies from 3.7 to 21.6% of adults depending on the population studied (country and age class), the method of diagnosis and the definition adopted. In the absence of available data for France, we analyzed the prevalence of Fuchs Endothelial Corneal Dystrophy (FECD) in a specific sub-population.

DETAILED DESCRIPTION:
The Primary purpose is to Estimate the prevalence of Fuchs' endothelial dystrophy in the French population in dermatology population.

ELIGIBILITY:
Inclusion Criteria:

* Patient with screening of Fuchs endothelial corneal dystrophy

Exclusion Criteria:

* Patients under guardianship
* Patients unable to receive informed consent
* Patients with anterior segment pathology (declarative) (the eye concerned will not be photographed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with screening of Fuchs endothelial corneal dystrophy will be included.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Dark spot in specular microscopy | Years: 1
  Dark sport or guttae after specular microscopy in parallel with the dermatological consultation

SECONDARY OUTCOMES:
Prevalence of Fuchs endothelial corneal dystrophy (FECD) as a function of age | Years: 1
  Prevalence of Fuchs endothelial corneal dystrophy (FECD) as a function of age. Data of medical record will be analyzed.
Prevalence of Fuchs endothelial corneal dystrophy (FECD) as a function of gender | Years: 1
  Prevalence of Fuchs endothelial corneal dystrophy (FECD) as a function of gender.
  Data of medical record will be analyzed.
Correlation between Fuchs endothelial corneal dystrophy (FECD) and skin pathology | Years: 1
  Correlation between Fuchs endothelial corneal dystrophy (FECD) and skin pathology.
  Data of medical record will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe GAIN, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No